CLINICAL TRIAL: NCT06083545
Title: The Effects of Application Intervention on the Physiological Indicators and Low Protein Diet Cognition Among the Patients With Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: yi ting Hsu (Other)
Responsible Party: Sponsor-Investigator, yi ting Hsu, nurse, Tri-Service General Hospital
Organization: Tri-Service General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ting652520
Record Dates: First submitted 2023-09-25; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: CKD Stage 4; CKD Stage 5
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Amyloid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: App — The low-protein diet app introduces the perceived significant efficacy of low-protein diets for patients with chronic kidney disease.
  Other Names: Application

SUMMARY:
The effects of Application intervention on the physiological indicators and low protein diet cognition among the patients with chronic kidney disease

DETAILED DESCRIPTION:
The low-protein diet app introduces the perceived significant efficacy of low-protein diets for patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or above and agree to participate in the research
* Conscious, literate and able to communicate in Mandarin and Taiwanese
* Have the ability to use vehicles
* Kidney disease stage is 3b as calculated by the MDRD formula From stage 5 to stage 5, he has not yet received alternative therapy and is diagnosed as a patient with chronic kidney disease by a nephrologist.

Exclusion Criteria:

* Blindness
* Cognitive abnormalities diagnosed by a doctor as dementia or mental disorder
* People who have no ability to act independently and are assisted by others in daily life
* Patients with nephrotic syndrome are excluded.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
basic information | 2 years
  Gender, age, education level, living status, financial resources, employment status, time of suffering from kidney disease, stage of kidney disease, time of nephrology treatment, combined chronic diseases, number of health education sessions by health teachers and nutritionists.
physiological index | 2 years
  It is an index for regular tracking and testing of research subjects. Information is provided by the laboratory department of the hospital of the research subjects. It mainly tracks serum potassium, phosphorus, sodium, calcium, and eGFR.
ow protein diet awareness scale | 2 years
  This scale was developed with reference to the Chronic Kidney Disease Health Management Manual of the Ministry of Health and Welfare (2018), with a total of 7 questions. It is scored as "true", "wrong" and "don't know", calculated on a scale of 0 to 1, with the highest It is 7 points, with forward and reverse questions. The higher the score, the more correct the understanding of low-protein diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Services General Hospital, Taipei, Neihu, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol